CLINICAL TRIAL: NCT02428205
Title: Combined Effects of Early Behavioral Intervention and Propranolol on ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Autism Science Foundation (Other)
Responsible Party: Principal Investigator, David Beversdorf, Associate Professor, Radiology, Neurology, Psychology, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2001935
Record Dates: First submitted 2015-04-16; First posted 2015-04-28 (Estimated); Results first posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propranolol arm (Experimental): Propranolol will be administered in the form of a liquid dose via oral syringe by the participants' parent/caregiver an hour before each EIBI session. To minimize risk, the bodyweight adjusted minimum dose of propranolol used safely for test anxiety in healthy adults (10mg) will be used: participants weighing > 30 kg will be given 4 mg, participants weighing 22.5 - 30 kg will be given 3 mg, participants weighing 15 - 22.5 kg will be given 2 mg. Participants weighing < 15 kg will be excluded for safety reasons.
  Interventions: Drug: Propranolol
- Placebo arm (Placebo Comparator): Placebo will be administered in the form of a liquid dose via oral syringe by the participants' parent/caregiver an hour before each EIBI session.The same bodyweight adjusted doses specified in the propranolol arm will be used for this arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — Participant will receive Propranolol prior to each EIBI session
  Other Names: Inderal
  Arms: Propranolol arm
Drug: Placebo — Participant will receive placebo prior to each EIBI session
  Arms: Placebo arm

SUMMARY:
The purpose of this study is to explore the effects of propranolol in combination with early intensive behavioral intervention on social interaction, and secondarily on language, anxiety, adaptive behaviors, and global function in children with autism in a double-blinded, placebo-controlled pilot trial.

DETAILED DESCRIPTION:
The investigators' specific aim is to examine the effects of serial doses of propranolol in combination with early intensive behavioral intervention on social interaction, and secondarily on language tasks, anxiety, adaptive behaviors, and global function in children with autism in a double-blinded, placebo-controlled trial. The investigators will also examine whether response to treatment can be predicted based upon markers of autonomic functioning, such as pupillary light reflex and heart rate variability, and whether anxiety predicts treatment response. The investigators' hypothesis is that propranolol will augment the effects of behavioral therapy on social functioning and language abilities. The investigators have demonstrated benefits of propranolol on social functioning and language in previous single-dose studies in adults and adolescents with autism. The investigators also predict that those with the greatest degree of autonomic dysregulation will demonstrate the greatest benefit from the drug.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism spectrum disorder (ASD), defined in this study by the DSM-V criteria plus Autism Diagnostic Observation Schedule (ADOS) criteria for Autism.
* Aged 3-8
* Participants must also be enrolled in an early behavioral intervention program at the Thompson Center or another institution in Missouri for the duration of the study.

Exclusion Criteria:

* Non-autism learning disability (e.g. dyslexia)
* Major psychiatric diagnosis (e.g. major depression, schizophrenia, bipolar disorder)
* Other neurological diagnosis
* Major head trauma
* Any of the following exclusionary criteria related to propranolol (diabetes, reactive airway/pulmonary disease, thyroid disease, bradyarrhythmias, unexplained syncope, narrow angle glaucoma, known hypersensitivity/adverse reaction to beta-blockers, potentially interacting drugs, underweight < 15 kg)
* Any of the following exclusionary criteria related to the use of electrocardiogram (history of rash from adhesives)
* Any of the following exclusionary criteria related to the pupillary reflex measurement (uncorrectable visual acuity impairment).
* Participants with a heart rate of less than 60 or a systolic blood pressure of less than 75 at the outset of the study will be excluded.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2015-04; Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Q Beversdorf, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- Thompson Center for Autism & Neurodevelopmental Disorders, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Allocated to Propranolol: Allocated to propranolol (n=5)
  Lost to follow-up (n=2)
  * Withdrew after baseline visit due to not feeling seeing a benefit (n=1)
  * Withdrew after 6-week visit -no reason given (n=1)
  Completed (n=4 at 6 weeks) (n=3 at 12 weeks)
- Allocated to Placebo: Allocated to placebo (n=4)
  Lost to follow-up (n=2)
  * Withdrew after baseline visit - no reason given (n=1)
  * Withdrew after baseline visit due to worsening behaviors (n=1)
  Completed (n=2 at 6 weeks) (n=2 at 12 weeks)
Period: Overall Study
Arm/Group | Allocated to Propranolol | Allocated to Placebo
Started | 5 | 4
Completed | 3 | 2
Not Completed | 2 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Worse behavior | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Propranolol Group: participants assigned to propranolol
- Placebo Group: participants assigned to placebo
- Total: Total of all reporting groups
Arm/Group | Propranolol Group | Placebo Group | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 4 | 9
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in General Social Outcome Measure (GSOM)
Description: The GSOM is a brief evaluation tool that measures a participant's level of social functioning and how it changes with intervention. There GSOM includes 4 different tasks: conversational reciprocity, ability to recognize facial expressions, social problem solving, affect demonstration, and emotional perspective taking. The experimenter administers each component of the GSOM to the participant and then scores their responses according to a pre-determined scoring rubric. Each component is scored on a 1-5 or 0 - 2 scale, with higher total scores indicating better social functioning. A video camera will be used to record the participant's behavior during GSOM administration for the purposes of having two independent raters score the tasks after the study session is complete. A camera will also be used during the affect demonstration task of the GSOM. The overall score is used. The range is 6-132, with higher scores being better.
Time Frame: Week 12
Population: This is a feasibility study so results are limited.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Propranolol Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
score on a scale | 48.3 (14.0) | 20.0 (15.6)

2. Primary Outcome: Change in Social Responsiveness Scale (SRS)
Description: This 65-item, parent-report measure asks questions about a participants' social awareness, social information processing, capacity for reciprocal social responses, social anxiety or avoidance, and characteristic autistic preoccupations or traits. The total score is used with a range of 0-195, with lower scores being better.
Time Frame: Week 12
Population: Feasibility only
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Propranolol Arm: Allocated to propranolol (n=5)
  Lost to follow-up (n=2)
  * Withdrew after baseline visit due to not feeling seeing a benefit (n=1)
  * Withdrew after 6-week visit -no reason given (n=1)
  Completed (n=4 at 6 weeks) (n=3 at 12 weeks)
- Placebo Arm: Allocated to placebo (n=4)
  Lost to follow-up (n=2)
  * Withdrew after baseline visit - no reason given (n=1)
  * Withdrew after baseline visit due to worsening behaviors (n=1)
  Completed (n=2 at 6 weeks) (n=2 at 12 weeks)
Arm/Group | Propranolol Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
score on a scale | 79.3 (17.0) | 72.0 (2.8)

3. Secondary Outcome: Change in Preschool Anxiety Scale (PAS)
Description: To assess anxiety, the PAS will be completed by the parents/caregivers of participants. This self-report measure yields a total score in addition to six subscales (separation anxiety, social phobia, obsessive compulsive, panic/agoraphobia, physical injury fears, and generalized anxiety). The overall score is used. Range is 0-112 with lower score meaning less anxiety.
Time Frame: Week 12
Population: Feasibility only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Propranolol Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
score on a scale | 87.7 (32.9) | 71.5 (30.4)

4. Secondary Outcome: Change in Aberrant Behavior Checklist (ABC)
Description: To assess overall behavioral disturbances, a parent/caregiver of the participants will complete ABC. This 58-item questionnaire is a well validated, reliable, and widely used assessment tool for interventions for a range of cognitive disorders. The full score is used, with a range of 0-174, with higher scores meaning more behaviors.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Propranolol Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
score on a scale | 72.7 (65.5) | 53.0 (39.6)

5. Secondary Outcome: Change in Vineland Adaptive Behavior Scales-II (VABS)
Description: To assess overall adaptive functioning, the VABS will be administered in the form of a structured interview with the parent/caregiver. The VABS is a well validated assessment used for the full range of our subjects' ages and yields standard scores in Communication, Daily Living Skills, Socialization, and Motor Skills. VABS scores for Socialization will be monitored in this study. The range is 20-160 with higher scores better.
Time Frame: Week 12
Population: Social domain
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Propranolol Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
score on a scale | 70.7 (10.2) | 66.5 (23.3)

6. Secondary Outcome: Change in Autism Impact Measure (AIM)
Description: The AIM will be administered to assess the frequency and impact of a participant's ASD-related symptoms. A parent/caregiver is asked a series of 41 questions regarding the frequency and the impact, or interference resulting from, a series of autism-associated behaviors. Peer interaction from the AIM is the primary domain obtained from this measure. For this domain the range is 0 to 40, with higher numbers more severe.
Time Frame: Week 12
Population: Peer interaction subdomain
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Propranolol Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
score on a scale | 23.7 (8.7) | 24.5 (6.4)

7. Secondary Outcome: Change in Preschool Language Scale (PLS):
Description: To evaluate language, we will administer the PLS, which has been developed for use in younger children (birth through age 7), and is appropriate for children of all ability levels, including nonverbal children. This play-based, interactive assessment is designed to assess receptive and expressive language skills and their change over time. The range is 50-150 with higher scores being better.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Propranolol Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
score on a scale | 87.7 (32.9) | 71.5 (30.4)

ADVERSE EVENTS:
Time Frame: Adverse event data collected for duration of medication administration- 12 weeks
Arm/Group | Propranolol Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 1/5 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propranolol Arm (N=5) | Placebo Arm (N=4)
Fatigue (General disorders) | 1 (1) | 0 (0) — Fatigue
aggression (General disorders) | 0 (0) | 1 (1) — aggression
irritability (General disorders) | 0 (0) | 1 (1) — irritability
insomina (General disorders) | 0 (0) | 1 (1) — insomnia

LIMITATIONS AND CAVEATS:
This was only a feasibility trial. We do not recommend emphasis be placed on the results due to the very small sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-19): https://cdn.clinicaltrials.gov/large-docs/05/NCT02428205/Prot_SAP_000.pdf